CLINICAL TRIAL: NCT03112187
Title: FLIPS: Ferfer Liposomal Iron Performance Study
Acronym: FLIPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PharmEvo Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PE/PK/FLIPS/SP/2017-01
Record Dates: First submitted 2017-03-27; First posted 2017-04-13 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-12

CONDITIONS: Iron Deficiency Anemia
Keywords: IDA; iron deficiency anemia; iron supplements; Pakistan; Liposomal iron
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Ferfer is a food supplement in liposomal form, with essential, vitamins including Vitamin C and Vitamin B12. Ferfer directly dissolves in the mouth without the need for water. The technology of liposomal microencapsulation, allows daily iron supplementation without any of the typical side effects of conventional oral iron supplements, such as heartburn, diarrhea, constipation, nausea and coloring of the mucous membranes and of the stools, which increases patient compliance. It has no metallic taste or smell, does not color mucous membrane and has excellent tolerability
  Interventions: Drug: Iron Supplement

INTERVENTIONS:
Drug: Iron Supplement — Ferfer® is a multi-ingredient supplement containing micro-encapsulated iron pyrophosphate (to form liposomes), vitamin C and vitamin B12 which are valuable for the control of nutritional deficiencies or increased organic needs of iron.
  Other Names: Micro liposomal iron

SUMMARY:
To evaluate the efficacy of a novel food supplement, Ferfer® to raise the capacity of Haemoglobin and Haematocrit levels

DETAILED DESCRIPTION:
Anemia, described as a low blood Haemoglobin concentration, has been shown to be a public health problem that impacts low-, center- and high-earnings nations and has great unfavorable health results, as well as unfavorable influences on social and monetary development . even though the most dependable indicator of anemia on the populace stage is blood Haemoglobin attention, measurements of this attention by myself do now not determine the cause of anemia. Anemia may additionally result from a number of causes, with the maximum great contributor being iron deficiency. approximately 30%- 50% of instances of anemia are taken into consideration to be because of iron deficiency.

Doctor will evaluate on the basis of inclusion or exclusion criteria, lab values and overall assessment and then enroll in this clinical trial. During the study patient will visit the Doctor four times, Day 0 week 4, week 8 and week 12. Doctor will investigate the Hemoglobin level and Hematocrit level and also evaluate the adverse effects and tolerability of Ferfer® at week 2 and week 8. Doctor also instructed to take the food supplements, twice daily, once in a morning and once in evening independently by food intake as Ferfer® has no interaction with food.

ELIGIBILITY:
Inclusion Criteria:

* Iron deficiency anemia (Hemoglobin <8 to >5 g/dl)
* Subjects able to provide written informed consent;
* Subjects already treated with other iron supplements or drugs that experienced side effects (not including allergy) related to iron administration.
* Wash out period will be a week

Exclusion Criteria:

* Had a history of iron intolerance
* Hypersensitivity and allergic of Vit C and Vit B12
* Not willing to take informed consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of a novel food supplement, Ferfer® to raise the capacity of Haemoglobin levels | Week 12
  To determine the efficacy of a novel food supplement,Ferfer® to raise the capacity of Haemoglobin levels
  Designated as safety issue: No

SECONDARY OUTCOMES:
Adverse Event | upto 12 weeks
  Number of Participants Who Experienced an Adverse Event
  [ Designated as safety issue: Yes ]
Efficacy of a novel food supplement, Ferfer® to raise the capacity of ferritin levels | Week 12
  To determine the efficacy of a novel food supplement, Ferfer® to raise the capacity of ferritin levels

CONTACTS AND LOCATIONS:
Overall Officials: Masood Jawaid, MRCS,FCPS, Study Director — PharmEvo Pvt Ltd
Locations (1):
- Lubna Shahzad,Al-raheem surgical and Maternity Hospital, Daroghwala, Lahore, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No